CLINICAL TRIAL: NCT05171413
Title: Predictive Models of Treatment Responses and Survival Outcomes in Patients With Soft Tissue Sarcoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuhan Yang, Associate Professor, West China Hospital
Other Study IDs: HX-20211156
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The internal cohort was retrospectively enrolled in West China Hospital, Sichuan University from June 2010 and December 2020. It is a training and internal validation cohort.
  Interventions: Other: Prediction model
- Prospective cohort: The same inclusion/exclusion criteria were applied for the same center prospectively. It is an external validation cohort.
  Interventions: Other: Prediction model

INTERVENTIONS:
Other: Prediction model — We develop and validate clinical models to predict treatment responses and survival outcomes in patients with biopsy-proven with soft tissue sarcoma.

SUMMARY:
The aim of this study was to developed and validated models to predict therapeutic responses and patients' survivals in patients with soft tissue sarcoma and compared these models with currently available models.

DETAILED DESCRIPTION:
We performed a retrospective-prospective cohort study with the aim of developing and validating comprehensive models to predict treatment responses and survival outcomes in patients with biopsy-proven soft tissue sarcoma. Secondly, we aimed to compare the predictive accuracy with currently available noninvasive model.

ELIGIBILITY:
Inclusion Criteria:

* Receiving no treatment before diagnosis
* With written informed consent

Exclusion Criteria:

* Clinical data missing
* Without written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with soft tissue sarcoma who were diagnosed histologically with definite pathologic specimens.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment response | At least 1-year follow up
  The primary outcome was the evaluation of treatment response to individualized therapy in patients with soft tissue sarcoma.
Progression-free survival outcomes | At least 5-year follow up
  The endpoint was defined as the occurrence of progression or recurrence, or the last follow-up. Patients were followed from the day of histological diagnosis until the occurrence of progression or recurrence, or last visit. The outcome was evaluated by an experienced oncologist in each center every 3-6 months. At each visit, a medical history, physical examination, and standard laboratory tests were performed.
Overall survival outcomes | At least 5-year follow up
  The endpoint was defined as the occurrence of death or the last follow-up. Patients were followed from the day of histological diagnosis until the occurrence of progression or recurrence or last visit. The outcome was evaluated by an experienced oncologist in each center every 3-6 months. At each visit, a medical history, physical examination, and standard laboratory tests were performed.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No